CLINICAL TRIAL: NCT05036590
Title: Efficiency Assessment of a Mental Health Professionals' Training Course for a Short Psychoeducational Program (BREF) for Families and Caregivers of Patients With Schizophrenia or First Psychotic Episode.
Brief Title: Efficiency Assessment of BREFORM. A Multicentric Stepped-wedge Randomized Control Trial.
Acronym: BREFORM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-A00269-30
Record Dates: First submitted 2021-08-05; First posted 2021-09-05 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Multicentric Stepped-wedge Randomized Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): The design is a stepped-wedge cluster randomized controlled trial. The study will be conducted in 9 centers (clusters) and will be conducted in 6 successive phases of 4 months each.
  During the first period, groups will be in the control period, then sequentially and according to a randomly defined order, at each time, one group will go into the intervention period after a transition period of 4 months allowing the intervention to be deployed (training of three health professionals for each center and then implementation of the BREF program).
  Thus, each cluster will belong successively to the control group and the intervention group. During the control period, caregivers will be supported according to the usual practices of each center. During the intervention period, the BREF program will be offered to all eligible caregivers.
  Interventions: Other: control group
- intervention group (Experimental): Thus, each cluster will belong successively to the control group and the intervention group. During the intervention period, the BREF program will be offered to all eligible caregivers.
  Interventions: Other: Intervention group

INTERVENTIONS:
Other: control group — The control group consisted of caregivers included during the control period, before the intervention was deployed, i.e., before the BREF program was implemented by the centers.
  Arms: Control group
Other: Intervention group — The intervention group consists of caregivers included during the intervention period. Caregivers in the intervention group will benefit from the BREF program.
  Arms: intervention group

SUMMARY:
In psychiatry, caregiver burden is associated with excess physical and psychological morbidity in relatives of patients with schizophrenic disorders Single or multi-family psychoeducation for caregivers of patients with schizophrenic disorders or first episode psychosis has a direct benefit on the health of the caregiver and an indirect benefit on the health of the ill family member. It is associated with a reduction in the rate of relapse and re-hospitalization and with better compliance with treatment. For single-family psychoeducation, the number of caregivers to be treated to avoid re-hospitalization of the sick family member is 3. For caregivers, psychoeducation is accompanied by an improvement in knowledge of the disorders and coping strategies. Therefore, international recommendations recommend that psychoeducation for caregivers be systematic, early, and integrated into routine care.

Currently, the organization of the French care system does not allow these recommendations to be met. In order to increase the use of psychoeducation in France, early interventions for caregivers must be offered systematically. The effectiveness of early psychoeducation for caregivers needs to be evaluated; only three randomized controlled trials are available in the literature and none have been conducted in France.

DETAILED DESCRIPTION:
The BREFORM project proposes to train health professionals in an early psychoeducation program, the BREF program, in order to implement it in their structure, and to evaluate its impact on the burden of caregivers of users living with a first psychotic episode or a schizophrenic disorder.

Regarding caregivers' outcomes:

outcome measures will be assessed at baseline (visit 1, V1), 6 weeks (Visit 2, V2), 6 months (Visit 3, V3), 12 months (Visit 4, V4) after baseline in the active group and in the treatment as usual group

Regarding patients' outcomes:

outcome measures will be assessed at baseline and 12 months after baseline in the active group and in the treatment as usual group

Regarding mental health professionals' outcomes:

outcome measures will be assessed before, after and 16 months after the training course

Regarding the psychiatric departments' outcomes:

outcome measures will be assessed at baseline and 36 months after baseline

ELIGIBILITY:
Inclusion Criteria:

* people over 18yo
* first-degree relatives (parents, siblings, children) or spouse of the patient
* primary caregiver of a patient with schizophrenic disorders or first psychotic episode (DSM5)
* consenting to participate to the study

Exclusion Criteria:

* mental disorder on Axis I
* having already benefited from a family intervention such as psychoeducation
* caring for several people with severe psychiatric disorders
* receiving income for the caring activities
* being legally responsible of the patient
* having difficulty understanding fluent French
* illiterate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2022-04-05 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the severity of caregiver burden between V1 and V4 by the Zarit Burden Inventory scale (ZBI) | one year
  The ZBI consists of 22 items rated on a 5-point Likert scale that ranges from 0 (never) to 4 (nearly always) with the sum of scores ranging between 0-88. Higher scores indicate greater burden. A score of 17 or more was considered high burden.

SECONDARY OUTCOMES:
Changes in caregiver burden severity at V1,V2 and V3 by the Zarit Burden Inventory (ZBI) scale | 8 months
  The ZBI consists of 22 items rated on a 5-point Likert scale that ranges from 0 (never) to 4 (nearly always) with the sum of scores ranging between 0-88. Higher scores indicate greater burden. A score of 17 or more was considered high burden.
Evolution of the caregivers' perceived-stress between V1, V2, V3, V4 by the Perceived Stress Scale-14 (PSS-14) | one year
  Total score of the PSS can be obtained by summing the 14 items' scores . The total score ranges from 0 to a maximum of 56, a higher score indicating a higher level of perceived stress.
Evolution of the caregivers' mood between V1, V2, V3, V4 by the Center for Epidemiologic Studies-Depression Scale (CES-D) | one year
  The CES-D consists of 20 items in a self-report format measuring depressive symptoms experienced in the past week on a 4-point Likert scale ranging from 0 (rarely or none of the time) to 3 (most or all of the time).
  Depression Severity: 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe. ... PHQ-9 score ≥10 had a sensitivity of 88% and a specificity of 88% for major depression.
Evolution of the caregivers' family functioning between V1, V2, V3, V4 | one year
  Assessed by the Family Assessment Device scale (FAD)
Evolution of the caregivers' quality of life between V1, V2, V3, V4 | one year
  Assessed by the Schizophrenia CareGiver Quality of Life scale (S-CGQoL)
Evolution of the caregivers' sense of competence between V1, V2, V3, V4 | one year
  assessed by the Sense of Competence Questionnaire scale (SCQ)
Evolution of the caregivers' number of consultations with the general practitioner (GP) | 12 months period before baseline assessment versus 12 months period after baseline assessment
  Change in number of consultations with the general practitioner (GP) n the 12 months prior to inclusion compared to the 12 months following inclusion
Evolution of the caregivers' number of days off work | 12 months period before baseline assessment vs. 12 months period after baseline assessment
  Change in number the caregivers' number of days off work in the 12 months prior to inclusion compared to the 12 months following inclusion
Evolution of the caregivers' number of days on long-term leave or disability | 12 months period before baseline assessment vs. 12 months period after baseline assessment
  Change in the number of long-term leaves of absence or disability related to the caregiver situation in the 12 months prior to inclusion compared to the 12 months following inclusion
Evolution of the caregivers' number of work days | 12 months
  Change in the number of work days related to the caregiver situation in the 12 months prior to inclusion compared to the 12 months following inclusion
Evolution of the caregivers' willingness to pay someone to replace them in their caring activities during one hour | 12 months
  Change in caregivers' willingness to pay someone to replace them in their caregiving activities for one hour in the 12 months prior to inclusion versus 12 months after inclusion.
Evolution of the caregivers' number of suicide attempts assessed by the Columbia Suicide Severity Rating Scale (C-SSRS) | 12 months period before baseline assessment vs. 12 months period after baseline assessment
  The Columbia Suicide Severity Rating Scale (C-SSRS) is a measure used to identify and assess individuals at risk for suicide. Questions are phrased for use in an interview format, but can be completed as a self-report measure if necessary.
  The score is created at each assessment for each patient and is used for determining treatment emergence. Suicidal Ideation Score: The maximum suicidal ideation category (1-5 on the C- SSRS) present at the assessment. Assign a score of 0 if no ideation is present.
caregivers' satisfaction | 12 months
  questionnaire
Evolution of the caregivers' living status (shared or non-shared household) between V1, V2, V3, V4 | 12 months
  questionnaire
Evolution of the caregivers' informal caregiving activities between V1, V2, V3, V4 | 12 months
  questionnaire
Evolution of the caregivers' number of hours spent providing informal caregiving between V1, V2, V3, V4 | 12 months
  questionnaire
Evolution of the patients' psychotic symptoms severity between baseline and 12 months after baseline assessed by the Positive And Negative Syndrome Scale (PANSS) | 12 months period before baseline assessment vs. 12 months period after baseline assessment
  PANSS items are rated on a 7-point scale (1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, and 7=extreme); because the absence of symptoms is equal to 1 point, the lowest possible total score on both PANSS scales is 7.
Evolution of the patients' functioning level between baseline and 12 months after baseline | Baseline assessment and 12 months after baseline assessment
  Assessed by the Global Assessment of Functionning scale (GAF)
Evolution of the patients' functioning level assessed by the Personal and social Performance scale (PSP) | Baseline assessment and 12 months after baseline assessment
  The patient's degree of severity in the four domains is to be rated on a six-point scale from absent (which means no problems on this dimension) over mild, manifest, marked, severe to very severe difficulties in the given area. Out of the ratings on the four subdimensions, one total score on a 100-point scale can be created. A variation of eight points is already to be classified as a clinically relevant difference. The items "self-care" and "disturbing and aggressive behavior" are of greater concern for patients with acute
Evolution of the patients' quality of life between baseline and 12 months after baseline | Baseline assessment and 12 months after baseline assessment
  Assessed by the Schizophrenia-quality of Life scale (S-QoL)
Evolution of the patients' clinical severity between baseline and 12 months after baseline | Baseline assessment and 12 months after baseline assessment
  Assessed by the Clinical Global Impression (CGI)
Evolution of the patients' depressive symptoms between baseline and 12 months after baseline | Baseline assessment and 12 months after baseline assessment
  Assessed by the Calgary Depression Scale for Schizophrenia scale (CDSS)
Evolution of the patients' relapse risk factors between baseline and 12 months after baseline | Baseline assessment and 12 months after baseline assessment
  Composite score assessed by the Medication Adherence Rating Scale (MARS) and Birchwood Scale (Birchwood), substance use disorders (declarative questionnaire)
Evolution of the patients' number of suicide attempts | 12 months period before baseline assessment vs. 12 months period after baseline assessment
  Assessed by the Columbia Suicide Severity Rating Scale " (C-SSRS)
Evolution of the patients' suicide risk level | Baseline assessment and 12 months after baseline assessment
  Assessed by the Columbia Suicide Severity Rating Scale " (C-SSRS)
Evolution of the patients' aggressive behaviors | 12 months period before baseline assessment vs. 12 months period after baseline assessment
  questionnaire
Evolution of the patients' number of hospitalization in psychiatry | 12 months period before baseline assessment vs. 12 months period after baseline assessment
  number of hospitalization in psychiatry
Evolution of the mental health professionals' beliefs and knowledge about psychoeducation to caregivers | Assessed before, after and 16 months after the training course
  questionnaire
Evolution of the mental health professionals' sense of competence about psychoeducation to caregivers | Assessed before, after and 16 months after the training course
  Self-assessment before, after and 16 months after the training course
Evolution of the mental health professionals' satisfaction of the training course | Assessed after and 16 months after the training course
  questionnaire
Evolution of the mental health professionals' satisfaction of the BREF program | Assessed 16 months after the training course
  questionnaire
Evolution of the psychiatric department organization regarding caregivers interventions | Assessed at baseline and 36 months after baseline
  questionnaire
Sustainability of the BREF program in each psychiatric department | Assessed 36 months after baseline
  Question the referent person at the center to know if the program is still used 3 years after its implementation
  QUESTION THE REFERENT PERSON AT THE CENTER TO KNOW IF THE PROGRAM IS STILL USED 3 YEARS AFTER ITS IMPLEMENTATION
  Question the referent perso of the center to know if the program is still used 3 years after its implementation

CONTACTS AND LOCATIONS:
Overall Officials: Romain REY, MD, PhD, Principal Investigator — CH LE VINATIER
Locations (1):
- Hopital Vinatier, Bron, France

IPD SHARING:
Plan to Share IPD: Undecided